CLINICAL TRIAL: NCT06064552
Title: Screening For First Trimester's Hyperglycemia in High and Low Risk Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Ahmed Mohamed, resident at obstetric and gynacology department, Sohag University
Other Study IDs: soh-Med-23-09-04MS
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Screening for Hyperglycemia in First Trimester in High and Low Risk Pregnancy
MeSH Terms: interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high risk pregnancy: Pregnant women with history of gestational diabetes in previous pregnancies, Polycystic ovaries syndrome, history of Macrosomic baby in previous pregnancies, Past history of late third trimester fetal demise, Past history of polyhydramnios, Overweight /Obese women, Women diagnosed to have other endocrinopathies like suprarenal, thyroid or pituitary disorders, multi fetal pregnancies, Past history of shoulder dystocia, Past history of preeclampsia
  Interventions: Diagnostic Test: blood sugar
- low risk pregnancy: average risk population like primigravida healthy women or those with normal obstetric history.
  Interventions: Diagnostic Test: blood sugar

INTERVENTIONS:
Diagnostic Test: blood sugar — High and low risk women will undergo measuring fasting blood sugar after fasting 6-8hours with good hydration. then measuring blood sugar 1hrs and 2hrs postprandial. for patient with high results (FBS>95mg/dl, 1hr postprandial>126mg/dl, 2hrs postprandial >140mg/dl) should do HA1C if >5.6 consider it diabetic and dealing with whom positive as regard lifestyle management like diet and exercise 150 min. per week and whom not well controlled will be enrolled in pharmacological regimen as metformin.
  For whom measures normal will be tested by the same method at 20- 24 wks of gestation

SUMMARY:
Glucose intolerance is the commonest medical disorder complicating pregnancy. Hyperglycemia increases the risk of delivering a large for gestational age newborn (LGA) and related complications such as operative delivery, birth trauma and the poor adaptation of the newborn . Maternal risks of GDM include also polyhydramnios, preeclampsia, premature delivery, prolonged labor, uterine atony, postpartum hemorrhage, infection and progression of retinopathy which are the leading global causes of maternal morbidity and mortality .Detection of women at higher risk for GDM early in pregnancy is a desirable goal because interventions such as diet, medication, and exercise may be applied earlier in pregnancy and potentially can reduce later development of GDM or its associated morbidities. Most GDM cases are diagnosed after mid-gestation following an abnormal glucose challenge test (GCT). However, about 10% of patients with GDM can be diagnosed in the first trimester.

ELIGIBILITY:
Inclusion Criteria:

* • History of gestational diabetes in previous pregnancies

  * Polycystic ovaries syndrome
  * History of Macrosomic baby in previous pregnancies
  * Past history of late third trimester fetal demise
  * Past history of polyhydramnios
  * Overweight /Obese women Women diagnosed to have other endocrinopathies like suprarenal, thyroid or pituitary disorders Multi fetal pregnancies Past history of shoulder dystocia Past history of preeclampsia Family history of diabetes

In addition, a comparable group of low-risk women will be included like primigravida healthy women or those with normal obstetric history.

Exclusion Criteria:

* all patient not have thev inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: History of gestational diabetes in previous pregnancies
  * Polycystic ovaries syndrome
  * History of Macrosomic baby in previous pregnancies
  * Past history of late third trimester fetal demise
  * Past history of polyhydramnios
  * Overweight /Obese women Women diagnosed to have other endocrinopathies like suprarenal, thyroid or pituitary disorders Multi fetal pregnancies Past history of shoulder dystocia Past history of preeclampsia Family history of diabetes
  In addition, a comparable group of low-risk women will be included like primigravida healthy women or those with normal obstetric history.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-09-24 (Estimated); Study Completion 2024-09-24 (Estimated)

PRIMARY OUTCOMES:
blood sugar percentage | 1 year
  High and low risk women will undergo measuring fasting blood sugar after fasting 6-8hours with good hydration. then measuring blood sugar 1hrs and 2hrs postprandial. for patient with high results (FBS>95mg/dl, 1hr postprandial>126mg/dl, 2hrs postprandial >140mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He XJ, Qin FY, Hu CL, Zhu M, Tian CQ, Li L. Is gestational diabetes mellitus an independent risk factor for macrosomia: a meta-analysis? Arch Gynecol Obstet. 2015 Apr;291(4):729-35. doi: 10.1007/s00404-014-3545-5. Epub 2014 Nov 12. PMID 25388922
- [Background] Hadden DR, McLaughlin C. Normal and abnormal maternal metabolism during pregnancy. Semin Fetal Neonatal Med. 2009 Apr;14(2):66-71. doi: 10.1016/j.siny.2008.09.004. Epub 2008 Nov 4. PMID 18986856
- [Background] Auvinen AM, Luiro K, Jokelainen J, Jarvela I, Knip M, Auvinen J, Tapanainen JS. Type 1 and type 2 diabetes after gestational diabetes: a 23 year cohort study. Diabetologia. 2020 Oct;63(10):2123-2128. doi: 10.1007/s00125-020-05215-3. Epub 2020 Jul 29. PMID 32725280